CLINICAL TRIAL: NCT02877329
Title: Internet-delivered ACT for Treating the Psychological Effects of Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAS-IT_2009-0055_ACTHÖR
Record Dates: First submitted 2014-04-05; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Hearing Loss
Keywords: psychological effects
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-delivered ACT (Experimental): Guided Internet-delivered Acceptance and commitment therapy for 8 weeks
  Interventions: Behavioral: Internet-delivered ACT
- Wait list control (No Intervention): No treatment during 8 weeks

INTERVENTIONS:
Behavioral: Internet-delivered ACT — Therapist-guided Internet-delivered ACT (acceptance and commitment therapy) for 8 weeks
  Arms: Internet-delivered ACT

SUMMARY:
Randomized trial comparing internet-delivered ACT with therapist support against waiting list for persons with hearing loss and comorbid psychological distress

DETAILED DESCRIPTION:
Hearing loss is the most common sensory disability in the world. Hearing loss is an auditory disability which affects not only speech recognition, but also the ability to recognize, locate and identify sounds in one's environment. Today there are a variety of studies investigating the relationship between hearing loss and mental health. For example, there are studies showing that hearing loss can lead to depression, somatization, social isolation, worrying or anxiety, loneliness, smaller social networks, lower self-efficacy, sensitivity to stress, burnout, and impaired sleep quality and quality of life in comparison with people with normal hearing. Initial results from other studies indicate that acceptance may be of importance, as it in turn can lead to increased help-seeking.To avoid prolonged stress and a healthy self-efficacy could contribute to greater well-being of people with hearing loss. This is the first study to use ACT to improve psychological health in people with hearing loss through the process of psychological flexibility. The treatment is eight weeks long and internet delivered through self-help texts with weekly therapist support.

ELIGIBILITY:
Inclusion Criteria:

* HHIE-S score over 8
* Indication of comorbid psychological suffering/distress (defined as total score above 0 on PHQ9/GAD7 or below 1sd on QOLI)

Exclusion Criteria:

* No computer with internet connection
* Unability to understand written content
* Incomplete screening procedure
* A health condition that needs immediate care

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The Hearing Handicap Inventory for Elderly-Screening, change between pre and post treatment | through study completion, an average of 8 weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire Depression 9 (PHQ9), change between pre and post treatment | through study completion, an average of 8 weeks
Generalized Anxiety Disorder 7 (GAD7), change between pre and post treatment | through study completion, an average of 8 weeks
Quality of Life Inventory (QOLI), change between pre and post treatment | through study completion, an average of 8 weeks
Hearing Acceptance Questionnaire (HAQ), change between pre and post treatment | through study completion, an average of 8 weeks
Hearing Self-Efficacy (HSE), change between pre and post treatment | through study completion, an average of 8 weeks
Perceived Stress Scale-4 (PSS-4), change between pre and post treatment | through study completion, an average of 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Linköpings Universitet, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No